CLINICAL TRIAL: NCT04467099
Title: Prevalence of Flexor Hallucis Longus Tears, Associated Os Trigonum Excision, and Return to Play
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Forte Sports Medicine and Orthopedics (Other)
Responsible Party: Principal Investigator, David Porter, Orthopedic Surgeon, Forte Sports Medicine and Orthopedics
Other Study IDs: 1453238
Record Dates: First submitted 2020-06-17; First posted 2020-07-10 (Actual); Last update posted 2021-09-20 (Actual); Status verified 2021-09

CONDITIONS: Ankle Impingement; Tendon Tear
Keywords: flexor hallucis longus; os trigonum; return to play
MeSH Terms: interventions — X-Rays; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Os Trigonum Excision with Tear: Participants with flexor hallucis tendon tear
  Interventions: Other: Foot Exam Follow-Up; Radiation: X-ray; Other: Questionnaire
- Os Trigonum Excision without Tear: Participants without flexor hallucis tendon tear
  Interventions: Other: Foot Exam Follow-Up; Radiation: X-ray; Other: Questionnaire

INTERVENTIONS:
Other: Foot Exam Follow-Up — All participants will have a clinical assessment of their surgery foot by the study doctor.
Radiation: X-ray — Standard x-ray of the foot.
Other: Questionnaire — All participants will complete a questionnaire.

SUMMARY:
The study's aim is to determine the incidence of flexor hallucis tendon tears associated with os trigonum excision. The study will then compare the length until functional return to play of the patients who had flexor hallucis tendon tears with concomitant os trigonum excision versus those without flexor hallucis tendon tears who underwent os trigonum excision. Lastly, the study will be evaluating the patient complaints and physical exam findings before and after surgery and compare those without flexor hallucis tendon tears to those with flexor hallucis tendon repair.

DETAILED DESCRIPTION:
Posterior ankle pain syndrome has many etiologies. Two main causes of this are flexor hallucis tendon tear and os trigonum impingement. The current teaching is that patients with flexor hallucis longus tear complain of posterior medial ankle pain and those with posterior lateral ankle pain have an os trigonum impingement. It is also classically understood that patients with flexor hallucis tendon tears take longer to return to their pre-injury level of function. Our clinical experience refutes these reports and our study looks to further evaluate it.

This study brings back patients who were treated by the study doctor. The patient's preoperative evaluation will be reviewed including clinic notes and imaging. The operative reports for these patients will be reviewed to verify the surgery procedure performed. These patients will be included in the study and we will utilize the American Academy of Orthopedic Surgeons Foot, Ankle, and Lower Limb module that they have completed postoperatively. This measure of patient's functional and subjective satisfaction has already been completed by patients at their regularly scheduled follow up appointments and is available for review.

Prospectively, patients will be asked to return to the clinic for a follow-up evaluation, which includes a standard x-ray. All patients will be consented prior to data collection, minors included in this study will be asked to sign an assent as well. Many factors will be assessed such as; a range of motion test of the ankle utilizing goniometric technique, nerve path and function, stability ankle grading, radiologic findings, and patient-reported outcomes filled out pre and postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Os trigonum excision with or without a flexor hallucis longus tear in an athletic population (recreational to competitive)
* Males and females ages 11-50 at time of surgery

Exclusion Criteria:

* Any other injury that will affect their return to play or recovery process
* Individuals not actively involved in athletic sport/activity
* Pregnant women
* Any other concomitant injuries

Ages: 11 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Prior patients of the study doctor from August 1996 to June 2017 that underwent os trigonum excision and of the athletic population (recreational to competitive).
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-03-02 (Actual); Primary Completion 2022-08 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Incidence of flexor hallucis longus tears associated with os trigonum excision | Less than or equal to 30 days
  How many participants had a tear.

SECONDARY OUTCOMES:
Length until return to play | Less than or equal to 30 days
  Comparing the length until return to play of the patients who had flexor hallucis longus tears with concomitant os trigonum excision versus those without flexor hallucis longus tears who underwent os trigonum excision.
Patient responses to American Academy of Orthopaedic Surgeons (AAOS) Foot and Ankle questionnaire | preoperative; perioperative; intraoperative; Less than or equal to 30 days
  The questionnaire responses will be summarized and compared between os trigonum excision with a flexor hallucis longus tear and without a flexor hallucis longus tear groups using two-sample Student t-tests.
Patient responses to American Academy of Orthopaedic Surgeons (AAOS) Lower Limb questionnaire | preoperative; perioperative; intraoperative; Less than or equal to 30 days
  The questionnaire responses will be summarized and compared between os trigonum excision with a flexor hallucis longus tear and without a flexor hallucis longus tear groups using two-sample Student t-tests.
Change in foot and ankle nerve function | preoperative; perioperative; intraoperative; Less than or equal to 30 days
  The comparison includes but is not limited to patient nerve path and function. The findings will be summarized and compared between os trigonum excision with a flexor hallucis longus tear and without a flexor hallucis longus tear groups using chi-square tests or Fisher's exact tests.
Change in foot and ankle areas of pain | preoperative; perioperative; intraoperative; Less than or equal to 30 days
  The comparison includes but is not limited to posterior pain, plantarflexion pain, os trigonum resection site pain, and other areas of pain upon visit. The findings will be summarized and compared between trigonum excision with a flexor hallucis longus tear and without a flexor hallucis longus tear groups using chi-square tests or Fisher's exact tests.
Change in foot and ankle range of motion | preoperative; perioperative; intraoperative; Less than or equal to 30 days
  The comparison includes but is not limited to patient range of motion (ROM) test in degrees of the ankle by assessing plantarflexion, dorsiflexion, hindfoot angle, and subtalar motion. The findings will be summarized and compared between trigonum excision with a flexor hallucis longus tear and without a flexor hallucis longus tear groups using two-sample Student t-tests.
Change in foot and ankle stability | preoperative; perioperative; intraoperative; Less than or equal to 30 days
  The comparison includes but is not limited to patient range of motion (ROM) test of the ankle by assessing plantarflexion, dorsiflexion, hindfoot angle, and subtalar motion. The findings will be summarized and compared between trigonum excision with a flexor hallucis longus tear and without a flexor hallucis longus tear groups using chi-square tests or Fisher's exact tests.
Change in foot and ankle imaging for x-ray and magnetic resonance imaging | preoperative; perioperative; intraoperative; Less than or equal to 30 days
  The comparison includes but is not limited to how many patients have within and group differences in x-ray and magnetic resonance imaging (MRI). Changes to be compared will include but not limited to ankle alignment, os trigonum, the appearance of posterior talus, osteochondral lesions, fractures or dislocations, stress fractures, plantar and posterior heel spurs and arthritic changes in the ankle or hindfoot.

CONTACTS AND LOCATIONS:
Overall Officials: David Porter, MD, PhD, Principal Investigator — Forte Sports Medicine and Orthopedics
Locations (2):
- United States (2):
  - Methodist Sports Medicine Carmel, Carmel, Indiana
  - Methodist Sports Medicine Greenwood, Greenwood, Indiana

IPD SHARING:
Plan to Share IPD: Undecided